CLINICAL TRIAL: NCT07066449
Title: Clinical Performance Evaluation of the Vivid Pioneer Diagnostic Ultrasound System
Brief Title: Clinical Performance Evaluation of a Diagnostic Ultrasound System
Status: Recruiting | Type: Observational
Sponsor: GE Healthcare (Industry)
Responsible Party: Principal Investigator, Juan Zhang, Deputy Chief Physician, Nanjing First Hospital, Nanjing Medical University
Other Study IDs: KY20250225-05
Record Dates: First submitted 2025-03-12; First posted 2025-07-15 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Echocardiography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Subjects who are required to undergo transesophageal echocardiography according to the current clinical practice standards will be eligible for enrollment. Subjects will be screened for enrollment in this study against the inclusion and exclusion criteria. After successful screening and enrollment of subjects, the investigators will first use the investigational device to conduct transthoracic echocardiography (TTE), followed by transesophageal echocardiography (TEE). TEE will be conducted after the subject has been anesthetized. To avoid any delay in diagnosis and treatment, after the scan with the investigational device is completed, the probe will be reserved and the console will be switched to the existing commercial cardiac diagnostic ultrasound device in the study site for intraoperative guidance. In the study, each investigator will evaluate the overall image quality, user interface, workflow, user preferences, product preset, and functions of the system, as well as the device's safety and stability and fill out a user feedback questionnaire provided by the Sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 18 years old, have autonomous capacity;
2. Subjects who are required to undergo intraoperative transesophageal echocardiography according to the current clinical practice standards;
3. Agree to participate in this study and have signed the subject Informed Consent Form.

Exclusion Criteria:

1. Subjects who have been previously enrolled in this study or are participating in other clinical trials;
2. Subjects with any medical emergency condition requiring urgent treatment;
3. Pregnant females;
4. Subjects with absolute contraindications of TEE (congenital or acquired upper digestive tract diseases, such as active upper gastrointestinal hemorrhage, esophageal obstruction or stenosis, esophageal tumor, esophageal lacerations and perforations, esophageal diverticula) or relative contraindications (changes in consciousness or lack of cooperation, history of cervical and mediastinal radiotherapy, history of recent esophageal surgery, esophageal varicosity, clotting disorders, cervical disease and injury, active esophagitis, active gastrointestinal ulcers, hiatal hernia, poor cardiopulmonary function, airway damage, pharyngeal space-occupying lesions, etc.), who are expected to be at high risks;
5. Any other subjects who should not participate in this study in the investigator's opinion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are required to undergo intraoperative transesophageal echocardiography according to the current clinical practice standards;
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
The main evaluation indicators include Overall system operation, Reliability, System operability, Overall image quality, etc., and the evaluation results are represented by five grades: Excellent, Very good, Good, Bad, and Very bad. | From enrollment to Day 1 （Visit 1）

OTHER OUTCOMES:
The other evaluation indicators include Imaging Mode , Structural Heart Disease Workflow Productivity Tools, FlexiSlice Improvements , The results are expressed as a score (5 to 1 point), with higher scores indicating better performance | From enrollment to Day1（Visit1）

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing First Hospital, Nanjing Medical University, Nanjing, China